CLINICAL TRIAL: NCT01625754
Title: The Heart-Mind Connection: Evaluating the Association Between Ceramides and Cognitive Decline in Coronary Artery Disease
Status: Completed | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Other Study IDs: 279-2011
Record Dates: First submitted 2012-05-24; First posted 2012-06-21 (Estimated); Last update posted 2024-01-31 (Actual); Status verified 2020-01

CONDITIONS: Coronary Artery Disease
Keywords: Ceramides; Lipids
MeSH Terms: conditions — Coronary Artery Disease | interventions — Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood for ApoE4 genotyping
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cardiac rehabilitation: This study recruits individuals that are currently participating in a cardiac rehabilitation exercise program.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — All individuals will be prescribed an exercise regimen according to their cardiac rehabilitation program

SUMMARY:
Many studies have shown that those with coronary artery disease (CAD) have a more rapid decline in memory than expected and that they are at an increased risk of developing dementia. It is not understood how memory decline is linked to CAD; however, it has recently been discovered that certain byproducts of fat breakdown involved in the development of CAD, called ceramides, can harm brain cells. In the present study the investigators will recruit 129 CAD patients from a cardiac rehabilitation facility and measure memory performance and blood ceramide concentrations at baseline, 3 months and 6 months. The investigators will also measure important blood messengers of inflammation and assess whether they are associated with ceramide production. In addition, relationships between ceramides and other aspects of brain function, such as thinking speed and the ability to plan and sort information will be explored.

DETAILED DESCRIPTION:
Coronary artery disease (CAD) affects about 19.8% of Canadians over the age of 65 and significantly affects quality of life. Of particular importance, cognitive impairment, ranging from cognitive complaints to vascular dementia, is frequently part of the clinical presentation of CAD. Our own prospective pilot data suggest that 22.5% of CAD patients attending cardiac rehabilitation (CR) have evidence of cognitive impairment with lower verbal memory performance, a marker of hippocampal function, predicting poorer CR outcomes. The pathophysiological mechanisms that may contribute to cognitive decline in those with CAD have not been fully elucidated.

Ceramides are metabolites of sphingomyelin, lipid species enriched in the outer leaflet of the plasma membrane and cell organelles of all tissues. Higher peripheral blood concentrations of ceramides have been associated with the development and progression of CAD. We propose to use a specific and sensitive electrospray ionization-tandem mass spectrometry (ESI-MS/MS) assay to measure concentrations of ceramide species from human plasma and elucidate the relationship between ceramides and the change in verbal memory performance over 6 months in 129 subjects with CAD undergoing CR.

We hypothesize that higher plasma concentrations of the long chain ceramide species C22:0 and C24:0 will be associated with decline in verbal memory performance and overall cognitive performance as assessed by a standardized battery of cognitive tests recommended for the investigation of vascular cognitive impairment. We also hypothesize that changes in the plasma concentration of TNF-α (tumor necrosis factor-alpha) will be associated with changes in plasma concentrations of C22:0 and C24:0 over 6 months.

This study aims to clarify the significance of a novel mechanism involving ceramides and the propagation of inflammatory signals from the periphery to the brain in mediating neurodegeneration associated with CAD.

ELIGIBILITY:
Inclusion Criteria:

* 50-75 years of age
* speak and understand English
* evidence of CAD based on at least 1 of the following:
* previous hospitalization for myocardial infarction
* angiographic evidence of ≥ 50% blockage in ≥ 1 major coronary artery
* a prior revascularization procedure
* no recent (last 4 weeks) hospitalization for cardiac events such as acute myocardial infarction, unstable angina, congestive heart failure, ventricular arrhythmias, coronary revascularization, or Canadian Cardiovascular Society Class 4 angina

Exclusion Criteria:

* Type I diabetes
* hypothyroidism, Parkinson's disease, any diagnosis of dementia including Alzheimer's disease, inflammatory disease (irritable bowel syndrome, Crohn's, arthritis, etc.), Huntington's chorea, brain tumour, other conditions that may affect cognitive performance such as history of epilepsy, subdural hematoma, traumatic brain injury, and clinical stroke, progressive supranuclear paralysis, Killip Class III or IV states, multiple sclerosis, severely disrupted liver/ kidney/ lung function
* use of hypnotics, antipsychotics, antidepressants, and anticholinergic medication
* premorbid psychiatric diagnosis of schizophrenia or bipolar disorder
* significant cognitive impairment (MMSE ≤ 24)
* diagnosis of any current Axis I disorder other than depression, phobias or nicotine abuse/dependence

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with coronary artery disease participating in a cardiac rehabilitation exercise program
Sampling Method: Probability Sample
Enrollment: 129 (Estimated)
Dates: Start 2011-11; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Change in Verbal memory | 6 months
  Verbal memory will be assessed using the California Verbal Learning Test, 2nd Edition (CVLT-II)

SECONDARY OUTCOMES:
Neuropsychiatric battery | Baseline, 3 months, 6 months
  The neuropsychiatric assessment battery recommended by the National Institute of Neurological Disorders and Stroke and the Canadian Stroke Network (NINDS-CSN) harmonized standards will be conducted
Montreal Cognitive Assessment (MoCA) | Baseline, 3 months, 6 months
  The MoCA will be used to assess global cognition

CONTACTS AND LOCATIONS:
Overall Officials: Krista Lanctôt, PhD, Principal Investigator — Sunnybrook Health Sciences Centre; Nathan Herrmann, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Toronto Rehabilitation Institute - Cardiac Rehab, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chan P, Saleem M, Herrmann N, Mielke MM, Haughey NJ, Oh PI, Kiss A, Lanctot KL. Ceramide Accumulation Is Associated with Declining Verbal Memory in Coronary Artery Disease Patients: An Observational Study. J Alzheimers Dis. 2018;64(4):1235-1246. doi: 10.3233/JAD-180030. PMID 30010121
- [Result] Saleem M, Bandaru VV, Herrmann N, Swardfager W, Mielke MM, Oh PI, Shammi P, Kiss A, Haughey NJ, Rovinski R, Lanctot KL. Ceramides predict verbal memory performance in coronary artery disease patients undertaking exercise: a prospective cohort pilot study. BMC Geriatr. 2013 Dec 12;13:135. doi: 10.1186/1471-2318-13-135. PMID 24330446